CLINICAL TRIAL: NCT03234192
Title: A Randomized Clinical Controlled Study Comparing the Effectiveness of the Astym Technique, the Graston Technique, and Therapeutic Ultrasound in the Treatment of Lateral Epicondylosis.
Brief Title: Effectiveness of the Astym Technique, the Graston Technique, and Therapeutic Ultrasound in the Treatment of Lateral Epicondylosis.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruiting was halted due to methodology issues
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 16-02176
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Lateral Epicondylitis; Tennis Elbow; Posterolateral Rotator Instability
Keywords: extensor carpi radialis brevis; Therapeutic Ultrasound; Astym Treatment Technique; Graston Treatment Technique
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Therapeutic ultra sound (Active Comparator)
  Interventions: Procedure: Therapeutic ultra sound
- Astym Treatment Technique (Active Comparator)
  Interventions: Procedure: Astym Treatment Technique
- Graston Treatment Technique (Active Comparator)
  Interventions: Procedure: Graston Treatment Technique

INTERVENTIONS:
Procedure: Therapeutic ultra sound — This group will receive standard treatment consisting of eccentric strengthening, stretch, proximal strengthening, and education in addition to therapeutic ultra sound treatment.
  Arms: Therapeutic ultra sound
Procedure: Astym Treatment Technique — This group will receive standard treatment consisting of eccentric strengthening, stretch, proximal strengthening, and education in addition to Astym Treatment.
  Arms: Astym Treatment Technique
Procedure: Graston Treatment Technique — This group will receive standard treatment consisting of eccentric strengthening, stretch, proximal strengthening, and education in addition to Graston Treatment.
  Arms: Graston Treatment Technique

SUMMARY:
The purpose of this study is to examine the effectiveness of three common techniques for the treatment of lateral epicondylosis. Through objective and subjective assessments this study will determine the effectiveness of the Astym Treatment Technique, the Graston Treatment Technique, and therapeutic ultrasound in the conservative treatment of lateral epicondylosis. It is hypothesized that the more manual Astym technique and Graston technique will produce more significant results than the more frequently utilized ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Clients who are admitted to NYULMC Center for Musculoskeletal Care for outpatient occupational or physical therapy with a diagnosis of lateral epicondylosis will be included. To participate in the study participants must:
* Be able to follow a home exercise program
* Be able to consent to participation in the research study

Exclusion Criteria:

* Clients who are deemed unable to consent to participation in the research study and/or unable to following a home exercise program will not be included in this study
* Clients with additional acute orthopedic injuries and/or surgeries to the involved upper extremity will not be included in this study.
* Clients with open wounds of the involved upper extremity that will interfere with treatment techniques will not be involved in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-06-10 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Patient Rated Tennis Elbow Evaluation (PRTEE) | 30 Minutes
  This is a 15 item self-reported questionnaire to measure perceived pain and disability in people with Lateral Epicondylosis (LE)
QuickDASH | 30 Minutes
  This is an 11 item questionnaire where by participants' score themselves using a 1-5 point scale. 1 represents "no difficulty" in performing task whereas 5 represents "unable to perform task"

SECONDARY OUTCOMES:
EQ-5D-5L | 30 Minutes
  This is a visual analog scale used to assess the clients view of their overall health on a scale of 0 (worst imaginable) to 100 (best imaginable). Also, clients report issues with mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each is scored on a 3 point scale.
Range of motion | 30 Minutes
  This will be taken at the wrist and elbow using goniometric measurements and a volar/dorsal approach at the wrist and lateral approach at the elbow. Measurements recorded will be wrist flexion and extension and elbow flexion and extension
Grip strength | 30 Minutes
  This will be measured using a hand held dynamometer and tested in the standard (arm at side) position and elbow extension position. Three trials on each UE will be reported in pounds
Numeric Rating Scale for Pain | 30 Minutes
  This scale is a single point scale from 0-10. The client picks one number to represent their pain, where 0 represents no pain and 10 represents worst pain imaginable
Cozens Test | 30 Minutes
  This involves the examiner resisting the wrist extension force of the client with the elbow in extension
Mills Test | 30 Minutes
  This is performed by palpating the lateral epicondyle while passively pronating the forearm, flexing the wrist, and extending the elbow

CONTACTS AND LOCATIONS:
Overall Officials: Steve Vanlew, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data.